CLINICAL TRIAL: NCT02125903
Title: Randomized Controlled Study: Comparison of Continuous Femoral Nerve Block and Adductor Canal Block After Total Knee Replacement Therapy Relating to Early Mobilization and Analgesia
Brief Title: Comparison of Continuous Femoral Nerve Block and Adductor Canal Block After Total Knee Replacement Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Karolin Piechowiak, Dr. Karolin Piechowiak, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AZ 06/13
Record Dates: First submitted 2014-02-05; First posted 2014-04-29 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Total Knee Arthroplasty; Total Knee Replacement; Femoral Nerve Block; Adductor Canal Block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Adductor Canal Block (CACB) (Active Comparator): Continuous Adductor Canal block performed with:
  loading dose 0,375% Ropivacaine 15ml (56,25mg) start infusion 0,2% Ropivacaine 6ml/h
  Procedure: Femoral Nerve Block. Adductor Canal Block Drug: Ropivacaine
  Interventions: Drug: Ropivacaine
- Continuous Femoral Nerve Block (CFNB) (Active Comparator): Continuous Femoral Nerve Block performed with:
  loading dose 0,375% Ropivacaine 15ml (56,25mg) start infusion 0,2% Ropivacaine 6ml/h
  Procedure: Femoral Nerve Block. Adductor Canal Block Drug: Ropivacaine
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Regional Anesthesia performed with 0.375% Ropivacaine 15ml (56,25mg)

SUMMARY:
The blockade of the femoral nerve (FNB) is the most common postoperative pain therapy after total knee replacement. Because of motor-driven weakness of the quadriceps muscle induced by femoral nerve block mobilization of Patients is difficult even dangerous (falls) and hospital stays are extended.

An alternative method could be an adductor canal block (ACB). Anatomical studies of the adductor canal demonstrated that the adductor canal contains the saphenous nerve, a pure sensory nerve for medial and anterior aspects of the knee and the tibia without any motor function.

This prospective, double-blinded, randomized study investigates the effect of FNB and ACB on quadriceps motor weakness and analgesia determined by Numeric Rating Scale (NRS).

We expect the ACB to be superior in muscle strength but equal in pain score. Both groups receive an additional anterior sciatic nerve block for complete sensory block of the operated knee

ELIGIBILITY:
Inclusion Criteria:

* patients with knee replacement therapy and general anaesthesia
* informed consent
* preoperative "timed up and go" test performable

Exclusion Criteria:

* emergency patients
* BMI > 40 kg/m2
* American Society of Anaesthesiologists physical status (ASA) 4-5
* severe chronic obstructive pulmonary disease (COPD)
* rheumatic arthritis, diabetic Polyneuropathy, M. Parkinson
* nerve injury of lumbosacral plexus
* coagulopathy with bleeding tendency
* not capable of speaking or understanding german or english

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Timed-Up and Go-test for mobility evaluation | third postoperative day
  The patient is observed and timed while he rises from an arm chair, walks 3 meters, turns, walks back, and sits down again.

SECONDARY OUTCOMES:
Pain Scores | 6, 24, 48, 72 hours postoperative
  Numeric Rating Scale (NRS), 0-10 for Rest / Stress. in Addition total Body NRS Pain
Quadriceps strength | 6, 24, 28, 72 hours postoperative
  Numeric Scale (0-5)
Ropivacaine consumption (each catheter) | 24, 48, 72 hours postoperative
  Measurement of the total amount
CAS (Cumulated Ambulation Score) | 24,48,72 hours postoperative
  Cumulated Ambulation Score is calculated with routine data. Measurement for ambulation ability
Mobility Score (MoSc) | 24,48,72 hours postoperative
  Is calculated with routine data. Measurement for overall mobilization (none- passive mobilization, sitting, standing, walking with walking device, walkin free or with crutches)
Analgesic regimen | preop and 0, 6 , 24, 48, 48 hours postoperative
  Documentation of analgesic prescriptions and rescue medications during postoperative course

CONTACTS AND LOCATIONS:
Overall Officials: Karolin Piechowiak, Dr, Study Director — Dept. of Anesthesia And Intensiv Care Medicine University of Marburg; Thorsten Steinfeldt, Prof Dr, Study Director — Dept. of Anesthesia And Intensive Care Medicine University of Marburg; Thomas Wiesmann, Dr, Study Director — Dept. of Anesthesia And Intensive Care Medicine University of Marburg
Locations (1):
- University of Marburg Department of Anaesthesia And Intensive Care Medicine, Marburg, Germany